CLINICAL TRIAL: NCT03317704
Title: Regulation of Metabolism and Ion Handling - Effect of High Intensity Training and NAC-infusion in Young Men
Brief Title: Regulation of Metabolism and Ion Handling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morten Hostrup, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Hostrup, PhD, Assistant Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SET-NAC
Record Dates: First submitted 2017-10-03; First posted 2017-10-23 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- speed endurance training (SET) (Active Comparator): Training 6 weeks 3 times pr. week
  Interventions: Behavioral: Speed endurance training
- Controls (No Intervention): Asked to continue their usual life style
- speed endurance training (SET) II (Active Comparator): Training 6 weeks 3 times pr. week
  Interventions: Behavioral: Speed endurance training

INTERVENTIONS:
Behavioral: Speed endurance training — Speed endurance training
  Arms: speed endurance training (SET); speed endurance training (SET) II

SUMMARY:
This study investigates the relation between ion-handling (K+) and fatigue development during exercise. Before and after a 6-week period of high intensity interval training, performance and ion-handling is assessed in young adults. In addition, mitochondrial function is examined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* 45-55 ml/kg/min
* BMI 19-26 kg/m2
* Normal ECG (assessed by MD)

Exclusion Criteria:

* Allergic to n-acetylcystine (NAC) or digoxin
* Severe side effects from NAC or digoxin
* Chronic diseases (assessed by MD to be a potential hazard or to interfere with outcome measures)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Quadriceps endurance | Change from before (baseline) to after 6 weeks of training (Week 6)
  Time to exhaustion during knee-extensor exercise

SECONDARY OUTCOMES:
K+ release | Change from before (baseline) to after 6 weeks of training (Week 6)
  Net leg K+ release in mmol/min during knee-extensor exercise

OTHER OUTCOMES:
Femoral venous plasma K+ | Change from before (baseline) to after 6 weeks of training (Week 6)
  Femoral venous plasma K+ in mmol/L during knee-extensor exercise
Femoral venous lactate | Change from before (baseline) to after 6 weeks of training (Week 6)
  Femoral venous lactate in mmol/L during knee-extensor exercise
Muscle Na+/K+-ATPase subunit content | Change from before (baseline) to after 6 weeks of training (Week 6)
  Muscle Na+/K+-ATPase subunit content from vastus lateralis biopsies
Muscle mitochondrial respiration | Change from before (baseline) to after 6 weeks of training (Week 6)
  Muscle mitochondrial respiration by high resolution respirometry (flux per mg muscle) from vastus lateralis biopsies
Muscle mitochondrial content | Change from before (baseline) to after 6 weeks of training (Week 6)
  Muscle mitochondrial content of citrate synthase from vastus lateralis biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided